CLINICAL TRIAL: NCT03290716
Title: Diet, Exercise and Cardiovascular Health - Effect of Salt Substitute and Stepwise Salt Supply Control in Reducing Blood Pressure in the Elderly in Nursing Homes in China: a Factorial Cluster-randomized Controlled Trial
Brief Title: Diet, ExerCIse and carDiovascular hEalth (DECIDE) - Salt Reduction Strategies for the Elderly in Nursing Homes in China
Acronym: DECIDE-Salt
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University (Other)
Collaborators: Changzhi Medical College (Other); Xi'an Jiaotong University (Other); Hohhot Center for Disease Control and Prevention (Unknown); Yangcheng Ophthalmology Hospital (Unknown)
Responsible Party: Principal Investigator, Yangfeng Wu, Prof of Epidemiology and Sciences in Clincial Research, Peking University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2016YFC130020302
Record Dates: First submitted 2017-09-05; First posted 2017-09-25 (Actual); Last update posted 2021-06-11 (Actual); Status verified 2021-06

CONDITIONS: Blood Pressure

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- SS+SSSC (Experimental): Salt substitute plus stepwise salt supply control
  Interventions: Other: SS; Other: SSSC
- SS only (Experimental): Salt substitute only
  Interventions: Other: SS
- SSSC only (Experimental): Stepwise salt supply control only
  Interventions: Other: SSSC
- control (No Intervention): No salt substitute and no stepwise salt supply control

INTERVENTIONS:
Other: SS — Replace regular salt with market available potassium-enriched salt substitute in kitchens of nursing homes.
  Other Names: Salt substitution
  Arms: SS only; SS+SSSC
Other: SSSC — A stepwise approach to reduce salt used in the kitchen of nursing homes by controlling the supply of salt.
  Other Names: Stepwise salt supply control
  Arms: SS+SSSC; SSSC only

SUMMARY:
The DECIDE - Salt in Elderly (Diet, ExerCIse and carDiovascular hEalth - Salt Reduction Strategies for the Elderly in Nursing Homes in China) is to evaluate the effects, safety and cost-effectiveness of salt substitution (SS) and stepwise salt supply control (SSSC) in reducing blood pressure in Chinese elderly in nursing homes. The study will recruit over 960 old people from 48 nursing homes in northern China. The 48 nursing homes will be randomised into the following 4 groups.

1. salt substitute (SS) and stepwise salt supply control (SSSC);
2. SS only;
3. SSSC only; and
4. no SS and no SSSC (control).

The intervention will last over 2 years. The randomization will be conducted centrally after the baseline survey completed. Primary outcome will be the change in systolic blood pressure. The secondary outcomes include: the changes in diastolic blood pressure, 24hr urinary sodium, potassium and microalbumin, and incidence of hyperkalemia, hypokalemia, hyponatremia, cardiovascular events, and all causes death, and incremental cost-effectiveness ratio.

DETAILED DESCRIPTION:
The DECIDE - Salt in Elderly (Diet, ExerCIse and carDiovascular hEalth - Salt Reduction Strategies for the Elderly in Nursing Homes in China) is a study in the DECIDE project, which includes five studies. The others are DECIDE - Diet, DECIDE - Exercise, DECIDE - Obesity in Children, and DECIDE - Smart Living. The DECIDE - Salt in Elderly study is to evaluate the effects, safety and cost-effectiveness of salt substitution (SS) and kitchen-based stepwise salt supply control (SSSC) in reducing blood pressure in Chinese elderly in nursing homes. Specifically, the study aims include:

1. to test if a stepwise salt supply control strategy could significantly reduce systolic blood pressure among elderly living in nursing homes;
2. to test if replacing regular salt with the market available salt substitute could significantly reduce systolic blood pressure among elderly living in nursing homes; and
3. to test if the joint effect of the two strategies is larger than that from one of each.

The corresponding null hypotheses that will be tested are:

1. the mean change from the baseline in systolic blood pressure of elderly residents in nursing homes that are supplied with SS is equal to the mean change from the baseline in systolic blood pressure of elderly residents in nursing homes that are supplied with regular salt;
2. the mean change from the baseline in systolic blood pressure of elderly residents in nursing homes that apply SSSC is equal to the mean change from the baseline in systolic blood pressure of elderly residents in nursing homes that do not apply SSSC;
3. There is no interaction between the two interventions above.

The study will recruit over 960 old people from 48 nursing homes in northern China, where the mean salt intake is generally higher than 12 g/day. A 2x2 factorial cluster-randomized trial will be used to test two independent salt reduction strategies: 1) using salt substitute to replace the regular salt in the kitchen of nursing homes; and 2) training the nursing manager to control/reduce, step by step, the amount of salt supplied to the kitchen of nursing homes. The 48 nursing homes will be randomized to the following 4 groups.

1. salt substitute (SS) and stepwise salt supply control (SSSC);
2. SS only;
3. SSSC only; and
4. no SS and no SSSC (control).

A brief health education on salt and health will be applied to all four groups. The salt substitute (NaCl 62.5% and KCl 25%) will be centrally provided. And the Train-the-trainers model will be used to train the nursing home managers how to implement the SSSC.

The intervention will last over 2 years. The baseline examination including three blood pressure measurements and one 24-hr urine collection will be conducted for all participants. Fasting blood samples will be drawn for measurement of serum potassium and detect hyperkalemia, hypokalemia, hyponatremia and renal dysfunction.

The randomization will be conducted centrally by the study coordinating center at Peking University Clinical Research Institute, after the baseline survey completed.

All participants will be followed up for blood pressure measurements at 6, 12, 18 and 24 months, for serum potassium at 12 and 24 months, and for 24-hr urine collection at 24 months.

Study outcomes:

Primary outcome: The change in systolic blood pressure from baseline to follow-up.

Secondary outcomes: The incidence of hyponatremia, hyperkalemia, hypokalemia and renal dysfunction from the baseline to 24 months. The change in 24-hr urinary sodium, potassium and microalbumin from the baseline to 24 months. The change in diastolic blood pressure from baseline to follow-up. The incremental cost-effectiveness ratio (ICER). The incidence of cardiovascular events and all causes death during follow up.

Power analysis:

On the assumptions of a 20% dropout rate, an intraclass correlation of 0.02, the number of clusters of 48 and at least 20 elderly people in each nursing home, and an α value of 0.05, the study to detect a mean 3.0 mmHg reduction in systolic blood pressure (SD, 18 mm Hg) between the intervention groups would have a power of 0.81. To detect a 4.0 mmHg reduction in systolic blood pressure (SD, 18 mm Hg), the power of the same sample size would be 0.96.

Statistical analysis: Linear models adjusted for clustering based on participants with available measures were used to assess continuous outcomes. Frailty survival models that account for clustering based upon all randomised participants were used for analysis of the effects on cardiovascular and mortality outcomes. Generalized linear mixed model were used for analysis of effects on hyperkalemia, hypokalemia, hyponatremia and renal dysfunction..

Ethical considerations:

The study will be submitted to and approved by the Peking University IRB, which has the full accreditation from AAHRRP. The study salt substitute is the product available on Chinese market and has been approved manufactured according to the product standards issued by the ministry of health. The SSSC approach will take every step for 3 months and the biggest step of salt reduction will be just 10% of the original amount of use. And the study will ensure an interview will be conducted to collect the feedback before every next step will take place. The SSSC intervention will stop at any time that elderly people feel unlike the foods.

ELIGIBILITY:
Eligibility of nursing homes:

* To be eligible, the nursing home must has not participated in any salt reduction or other intervention trials, has at least 20 residents and has agreed to participate in the study.

Eligibility of individual elderly:

Inclusion Criteria:

* Living in the nursing home permanently or expectedly for the coming two years
* Age less than 55 years.
* Life expectancy over six months.
* Provide written informed content.

Exclusion Criteria:

* Clinically confirmed hyperkalemia

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1612 (Actual)
Dates: Start 2017-09-25 (Actual); Primary Completion 2020-10-24 (Actual); Study Completion 2021-05-11 (Actual)

PRIMARY OUTCOMES:
The change in systolic blood pressure from baseline to follow-up | baseline、6 month、12 month、18 month and 24-month follow-up
  mmHg

SECONDARY OUTCOMES:
The incidence of hyperkalemia | throughout 24 months of follow-up
  A new case of hyperkalemia is defined as having serum potassium >5.5 mmol/L at either month 12 or 24 among participants with normal serum potassium at the baseline, regardless of clinical manifestations.
The incidence of hypokalemia | throughout 24 months of follow-up
  A new case of hypokalemia is defined as having serum potassium <3.5 mmol/L at either month 12 or 24 among participants with normal serum potassium at the baseline, regardless of clinical manifestations.
The change in 24-hour urinary sodium and potassium | baseline and 24-month follow-up
  mmol/d
The change in 24-hour urinary microalbumin | baseline and 24-month follow-up
  mg/day
The change in diastolic blood pressure from baseline to follow-up | baseline、6 month、12 month、18 month and 24-month follow-up
  mmHg
ICER | throughout 24 months of follow-up
  Incremental cost-effectiveness ratio, defined by the difference in the cost for every unit of gain in the pertained effectiveness outcome
Cardiovascular events | throughout 24 months of follow-up
  fatal and nonfatal stroke, fatal and nonfatal myocardial infarction, hospitalization for congestive heart failure
Death | throughout 24 months of follow-up
  all causes death
The incidence of hyponatremia | throughout 24 months of follow-up
  A new case of hyponatremia is defined as having serum sodium <135 mmol/L at either 12 or 24 months with normal serum sodium at the baseline, regardless of clinical manifestations.
The incidence of renal dysfunction | throughout 24 months of follow-up
  A new case of renal dysfunction is defined as having eGFR <60 at either 12 or 24 months with normal eGFR at the baseline, regardless of clinical manifestations.

CONTACTS AND LOCATIONS:
Overall Officials: Yangfeng Wu, PhD, Principal Investigator — Peking University
Locations (1):
- Mishan Nursing Home, Jincheng, Shanxi, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhang X, Yuan Y, Li C, Feng X, Wang H, Qiao Q, Zhang R, Jin A, Li J, Li H, Wu Y. Effect of a Salt Substitute on Incidence of Hypertension and Hypotension Among Normotensive Adults. J Am Coll Cardiol. 2024 Feb 20;83(7):711-722. doi: 10.1016/j.jacc.2023.12.013. PMID 38355240
- [Derived] Lai X, Yuan Y, Wang H, Zhang R, Qiao Q, Feng X, Jin A, Li H, Li J, Si L, Gao P, Jan S, Fang H, Wu Y; DECIDE-Salt Research Group. Cost-Effectiveness of Salt Substitute and Salt Supply Restriction in Eldercare Facilities: The DECIDE-Salt Cluster Randomized Clinical Trial. JAMA Netw Open. 2024 Feb 5;7(2):e2355564. doi: 10.1001/jamanetworkopen.2023.55564. PMID 38345818
- [Derived] Yuan Y, Jin A, Zhao MH, Wang H, Feng X, Qiao Q, Zhang R, Gao R, Wu Y. Association of serum potassium level with dietary potassium intake in Chinese older adults: a multicentre, cross-sectional survey. BMJ Open. 2023 Nov 24;13(11):e077249. doi: 10.1136/bmjopen-2023-077249. PMID 38000815
- [Derived] Yuan Y, Jin A, Duan P, Cao L, Wang H, Hu S, Li J, Feng X, Qiao Q, Zhang H, Zhang R, Li H, Gao P, Xie G, Yuan J, Cheng L, Wang S, Niu W, Elliott P, Gao R, Labarthe D, Wu Y. Experience with 2 years' intervention to progressively reduce salt supply to kitchens in elderly care facilities-challenges and further research: post hoc analysis of the DECIDE-Salt randomized clinical trial. BMC Med. 2023 Nov 3;21(1):416. doi: 10.1186/s12916-023-03130-z. PMID 37919742
- [Derived] Yuan Y, Jin A, Neal B, Feng X, Qiao Q, Wang H, Zhang R, Li J, Duan P, Cao L, Zhang H, Hu S, Li H, Gao P, Xie G, Yuan J, Cheng L, Wang S, Zhang H, Niu W, Fang H, Zhao M, Gao R, Chen J, Elliott P, Labarthe D, Wu Y. Salt substitution and salt-supply restriction for lowering blood pressure in elderly care facilities: a cluster-randomized trial. Nat Med. 2023 Apr;29(4):973-981. doi: 10.1038/s41591-023-02286-8. Epub 2023 Apr 13. PMID 37055566
- [Derived] Jin A, Zhao M, Sun Y, Feng X, Zhang R, Qiao Q, Wang H, Yuan J, Wang Y, Cheng L, Zhang H, Li HJ, Wu Y. Normal range of serum potassium, prevalence of dyskalaemia and associated factors in Chinese older adults: a cross-sectional study. BMJ Open. 2020 Oct 30;10(10):e039472. doi: 10.1136/bmjopen-2020-039472. PMID 33127634